CLINICAL TRIAL: NCT00811395
Title: Long-term Extension of the Multinational, Double-blind, Placebo Controlled Studies PDY6045 and PDY6046 to Document the Safety of Teriflunomide When Added to Treatment With Interferon-Beta or Glatiramer Acetate in Patients With Multiple Sclerosis With Relapses
Brief Title: Long Term Safety of Teriflunomide When Added to Interferon-Beta or Glatiramer Acetate in Patients With Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LTS6047; HMR1726D/2005 (Other: HMR); 2007-003997-24 (EudraCT Number)
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Results first posted 2012-12-31 (Estimated); Last update posted 2012-12-31 (Estimated); Status verified 2012-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — teriflunomide; Interferon beta-1a; Interferon beta-1b; Glatiramer Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Placebo + IFN-β (Placebo Comparator): Placebo (for teriflunomide) once daily concomitantly with interferon-β [IFN-β] for 24 additional weeks
  Interventions: Drug: Placebo (for teriflunomide); Drug: Interferon-β [IFN-β]
- Teriflunomide 7 mg + IFN-β (Experimental): Teriflunomide 7 mg once daily concomitantly with interferon-β [IFN-β] for 24 additional weeks
  Interventions: Drug: Teriflunomide; Drug: Interferon-β [IFN-β]
- Teriflunomide 14 mg + IFN-β (Experimental): Teriflunomide 14 mg once daily concomitantly with interferon-β [IFN-β] for 24 additional weeks
  Interventions: Drug: Teriflunomide; Drug: Interferon-β [IFN-β]
- Placebo + GA (Placebo Comparator): Placebo (for teriflunomide) once daily concomitantly with glatiramer acetate [GA] for 24 additional weeks
  Interventions: Drug: Placebo (for teriflunomide); Drug: Glatiramer Acetate [GA]
- Teriflunomide 7 mg + GA (Experimental): Teriflunomide 7 mg once daily concomitantly with glatiramer acetate [GA] for 24 additional weeks
  Interventions: Drug: Teriflunomide; Drug: Glatiramer Acetate [GA]
- Teriflunomide 14 mg + GA (Experimental): Teriflunomide 14 mg once daily concomitantly with glatiramer acetate [GA] for 24 additional weeks
  Interventions: Drug: Teriflunomide; Drug: Glatiramer Acetate [GA]

INTERVENTIONS:
Drug: Teriflunomide — Film-coated tablet
  Oral administration
  Other Names: HMR1726
  Arms: Teriflunomide 14 mg + GA; Teriflunomide 14 mg + IFN-β; Teriflunomide 7 mg + GA; Teriflunomide 7 mg + IFN-β
Drug: Placebo (for teriflunomide) — Film-coated tablet
  Oral administration
  Arms: Placebo + GA; Placebo + IFN-β
Drug: Interferon-β [IFN-β] — Powder for reconstitution, of any licensed strength for either intramuscular or subcutaneous injection
  Other Names: Avonex®; Rebif®; Betaseron®
  Arms: Placebo + IFN-β; Teriflunomide 14 mg + IFN-β; Teriflunomide 7 mg + IFN-β
Drug: Glatiramer Acetate [GA] — Solution in prefilled syringe for subcutaneous injection
  Other Names: Copaxone®
  Arms: Placebo + GA; Teriflunomide 14 mg + GA; Teriflunomide 7 mg + GA

SUMMARY:
The primary objective was to evaluate the long-term safety and tolerability of teriflunomide when added to treatment with interferon-β [IFN-β] or glatiramer Acetate [GA] in patients with multiple sclerosis [MS] with relapses.

Secondary objectives were to evaluate the long-term effect on relapse rate, disability progression and Magnetic Resonance Imaging [MRI] parameters.

This study is the extension study of the PDY6045 (NCT00489489) and PDY6046 (NCT00475865) studies. Participants who successfully completed the initial study were offered to continue their treatment (same compound, same dose) for 24 additional weeks.

DETAILED DESCRIPTION:
The duration of the extension study per participants was 40 weeks broken down as follows:

* 24-week double-blind treatment period,
* 16-week post-treatment elimination follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* PDY6045 or PDY6046 participant who:

  * completed the week 24 visit of either study PDY6045 or PDY6046,
  * was still meeting eligibility criteria for receiving treatment,
  * had agreed to continue stable dose of Interferon-β [IFN-β] or Glatiramer Acetate [GA] and consented to continue on treatment.

Exclusion Criteria:

* Any known condition or circumstance that would have prevented in the investigator's opinion, compliance or completion of the study

The above information is not intended to contain all considerations relevant to patient's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 182 (Actual)
Dates: Start 2007-10; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (7):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Vienna, Austria
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Guildford, United Kingdom

REFERENCES:
- [Result] Freedman MS, Wolinsky JS, Wamil B, Confavreux C, Comi G, Kappos L, Olsson TP, Miller A, Benzerdjeb H, Li H, Simonson C, O'Connor PW; Teriflunomide Multiple Sclerosis Trial Group and the MRI Analysis Center. Teriflunomide added to interferon-beta in relapsing multiple sclerosis: a randomized phase II trial. Neurology. 2012 Jun 5;78(23):1877-85. doi: 10.1212/WNL.0b013e318258f7d4. Epub 2012 May 23. PMID 22622860
- [Derived] Freedman MS, Wolinsky JS, Truffinet P, Comi G, Kappos L, Miller AE, Olsson TP, Benamor M, Chambers S, O'Connor PW. A randomized trial of teriflunomide added to glatiramer acetate in relapsing multiple sclerosis. Mult Scler J Exp Transl Clin. 2015 Dec 7;1:2055217315618687. doi: 10.1177/2055217315618687. eCollection 2015 Jan-Dec. PMID 28607708

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 107 and 110 participants who successfully completed 24-week visit in, respectively, PDY6045 and PDY6046 studies, were offered to continue their treatment in this extension study.
  After signature of the informed consent and confirmation of selection criteria, 86 and 96 participants entered the extension study.
Pre-assignment Details: An Interactive Voice Response System was used to allocate kits containing the same treatment as in the initial study.
  Analysis included all participants randomized in the initial studies and all data collected from randomization according to intent-to-treat principal.
Groups:
- Placebo + IFN-β: Placebo (for teriflunomide) once daily concomitantly with interferon-β [IFN-β]
- Teriflunomide 7 mg + IFN-β: Teriflunomide 7 mg once daily concomitantly with interferon-β [IFN-β]
- Teriflunomide 14 mg + IFN-β: Teriflunomide 14 mg once daily concomitantly with interferon-β [IFN-β]
- Placebo + GA: Placebo (for teriflunomide) once daily concomitantly with Glatiramer Acetate [GA]
- Teriflunomide 7 mg + GA: Teriflunomide 7 mg once daily concomitantly with Glatiramer Acetate [GA]
- Teriflunomide 14 mg + GA: Teriflunomide 14 mg once daily concomitantly with Glatiramer Acetate [GA]
Period: Initial Treatment (PDY6045 or PDY6046)
Arm/Group | Placebo + IFN-β | Teriflunomide 7 mg + IFN-β | Teriflunomide 14 mg + IFN-β | Placebo + GA | Teriflunomide 7 mg + GA | Teriflunomide 14 mg + GA
Started | 41 | 37 (One participant received 7 mg instead of 14 mg as per randomization) | 38 | 40 | 42 | 41
Completed | 38 (completed 24-week treatment (for more information see PDY6045/NCT00489489 record)) | 33 (completed 24-week treatment (for more information see PDY6045/NCT00489489 record)) | 36 (completed 24-week treatment (for more information see PDY6045/NCT00489489 record)) | 38 (completed 24-week treatment (for more information see PDY6046/NCT00475865 record)) | 37 (completed 24-week treatment (for more information see PDY6046/NCT00475865 record)) | 35 (completed 24-week treatment (for more information see PDY6046/NCT00475865 record))
Not Completed | 3 | 4 | 2 | 2 | 5 | 6
Period: Extension Treatment
Arm/Group | Placebo + IFN-β | Teriflunomide 7 mg + IFN-β | Teriflunomide 14 mg + IFN-β | Placebo + GA | Teriflunomide 7 mg + GA | Teriflunomide 14 mg + GA
Started | 31 (continued initial treatment) | 28 (continued initial treatment) | 27 (continued initial treatment) | 37 (continued initial treatment) | 30 (continued initial treatment) | 29 (continued initial treatment)
Completed | 29 (completed 48-week treatment) | 22 (completed 48-week treatment) | 24 (completed 48-week treatment) | 34 (completed 48-week treatment) | 30 (completed 48-week treatment) | 27 (completed 48-week treatment)
Not Completed | 2 | 6 | 3 | 3 | 0 | 2
Not completed — Adverse Event | 1 | 2 | 2 | 2 | 0 | 1
Not completed — Progressive disease | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Participant did not wish to continue | 0 | 3 | 0 | 1 | 0 | 1
Not completed — Other than above | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + IFN-β | Teriflunomide 7 mg + IFN-β | Teriflunomide 14 mg + IFN-β | Placebo + GA | Teriflunomide 7 mg + GA | Teriflunomide 14 mg + GA | Total
Number analyzed (Participants) | 41 | 37 | 38 | 40 | 42 | 41 | 239
Age, Customized [Number; unit: participants] — Baseline characteristics before randomization in the initial study (PDY6045 or PDY6046)
  participants
    <38 years | 17 | 9 | 15 | 11 | 12 | 13 | 77
    >=38 years | 24 | 28 | 23 | 29 | 30 | 28 | 162
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 25 | 25 | 31 | 33 | 33 | 178
  Male | 10 | 12 | 13 | 9 | 9 | 8 | 61
Region of Enrollment [Number; unit: participants] — Europe: Austria, Germany, Italy, Spain and United Kingdom
  North America: Canada and United States
  participants
    Europe | 28 | 25 | 24 | 22 | 22 | 22 | 143
    North America | 13 | 12 | 14 | 18 | 20 | 19 | 96

OUTCOME MEASURES:

1. Primary Outcome: Overview of Adverse Events [AE]
Description: AE are any unfavorable and unintended sign, symptom, syndrome, or illness observed by the investigator or reported by the participant during the study.
Time Frame: from first study drug intake in PDY6045/PDY6046 study up to 112 days after last intake in initial study or in the extension study, whichever occured last (64 weeks max)
Population: All randomized and treated participants; Participants were included in the treatment group according to the drug actually received.
Measure: Number; unit: participants
Arm/Group | Placebo + IFN-β | Teriflunomide 7 mg + IFN-β | Teriflunomide 14 mg + IFN-β | Placebo + GA | Teriflunomide 7 mg + GA | Teriflunomide 14 mg + GA
Number analyzed (Participants) | 41 | 37 | 38 | 40 | 42 | 41
participants
  Any AE | 35 | 35 | 33 | 39 | 40 | 38
  - serious AE | 2 | 4 | 1 | 6 | 5 | 2
  - AE leading to death | 0 | 0 | 0 | 0 | 0 | 0
  - AE leading to study drug discontinuation | 2 | 3 | 3 | 2 | 3 | 5

2. Secondary Outcome: Annualized Relapse Rate [ARR]: Poisson Regression Estimates
Description: ARR is obtained from the total number of confirmed relapses that occured during the treatment period divided by the sum of the treatment durations.
  Each episode of relapse - appearance, or worsening of a clinical symptom that was stable for at least 30 days, that persisted for a minimum of 24 hours in the absence of fever - was to be confirmed by an increase in Expanded Disability Status Scale [EDSS] score or Functional System scores.
  To account for the different treatment durations among participants, two Poisson regression models with robust error variance were used (total number of confirmed relapses as response variable, log-transformed treatment duration as "offset" variable and:
  * Model 1 (IFN-β groups): treatment group, region of enrollment and IFN-β dose level as covariates
  * Model 2 (GA groups): treatment group and region of enrollment as covariates)
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: relapses per year
Arm/Group | Placebo + IFN-β | Teriflunomide 7 mg + IFN-β | Teriflunomide 14 mg + IFN-β | Placebo + GA | Teriflunomide 7 mg + GA | Teriflunomide 14 mg + GA
Number analyzed (Participants) | 41 | 37 | 38 | 41 | 42 | 40
relapses per year | 0.343 [0.162 to 0.727] | 0.231 [0.101 to 0.529] | 0.144 [0.065 to 0.318] | 0.420 [0.270 to 0.654] | 0.262 [0.140 to 0.489] | 0.497 [0.316 to 0.783]

3. Primary Outcome: Overview of AE With Potential Risk of Occurence
Description: AE with potential risk of occurrence were defined as follows:
  * Hepatic disorders;
  * Immune effects, mainly effects on bone marrow and infection;
  * Pancreatic disorders;
  * Malignancy;
  * Skin disorders, mainly hair loss and hair thinning;
  * Pulmonary disorders;
  * Hypertension;
  * Peripheral neuropathy;
  * Psychiatric disorders;
  * Hypersensitivity.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo + IFN-β | Teriflunomide 7 mg + IFN-β | Teriflunomide 14 mg + IFN-β | Placebo + GA | Teriflunomide 7 mg + GA | Teriflunomide 14 mg + GA
Number analyzed (Participants) | 41 | 37 | 38 | 40 | 42 | 41
participants
  Any AE with potential risk of occurence | 28 | 30 | 30 | 34 | 33 | 32
  - Hepatic disorder AE | 7 | 11 | 13 | 5 | 4 | 5
  - Immune effects related AE | 16 | 21 | 20 | 27 | 22 | 21
  - Pancreatic disorder AE | 8 | 5 | 11 | 6 | 6 | 11
  - Malignancy AE | 0 | 0 | 0 | 0 | 0 | 0
  - Hair loss / hair thinning AE | 1 | 3 | 4 | 1 | 5 | 7
  - Pulmonary disorder AE | 0 | 0 | 0 | 0 | 1 | 0
  - Hypertension-related AE | 1 | 4 | 6 | 0 | 2 | 2
  - Peripheral neuropathy AE | 5 | 3 | 4 | 4 | 5 | 10
  - Psychiatric disorder AE | 1 | 1 | 2 | 3 | 3 | 1
  - Hypersensitivity AE | 6 | 4 | 4 | 4 | 6 | 10

4. Secondary Outcome: Overview of 12-week Sustained Disability Progression
Description: 12-week sustained disability progression was defined as an increase from baseline of at least 1-point in EDSS score (at least 0.5-point for participants with baseline EDSS score >5.5) that persisted for at least 12 weeks.
  If no disability progression was observed on or before last EDSS evaluation before study drug discontinuation, then the participant was considered as free of disability progression.
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo + IFN-β | Teriflunomide 7 mg + IFN-β | Teriflunomide 14 mg + IFN-β | Placebo + GA | Teriflunomide 7 mg + GA | Teriflunomide 14 mg + GA
Number analyzed (Participants) | 41 | 37 | 38 | 41 | 42 | 40
participants
  Disability progression | 0 [0.0 to 0.0] | 3 [0.0 to 8.9] | 2 [0.0 to 7.9] | 4 [0.0 to 7.3] | 1 [0.0 to 0.0] | 4 [0.0 to 13.2]
  Free of disability progression | 40 [0.0 to 0.0] | 33 [0.00 to 23.1] | 36 [0.0 to 15.2] | 37 [0.7 to 20.4] | 41 [0.0 to 9.8] | 36 [1.0 to 24.6]

5. Secondary Outcome: Time to 12-week Sustained Disability Progression: Kaplan-Meier Estimates of the Rate of Disability Progression at Timepoints
Description: Probability of disability progression at 24 and 48 weeks was estimated using Kaplan-Meier method on the time to disability progression defined as the time from randomization to first EDSS increase. Participants free of disability progression were censored at the date of the last on-treatment EDSS evaluation.
  Kaplan-Meier method consists in computing probabilities of non occurrence of event at any observed time of event and multiplying successive probabilities for time ≤t by any earlier computed probabilities to estimate the probability of being event-free for the amount of time t. Probability of event at time t is 1 minus the probability of being event-free for the amount of time t.
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Placebo + IFN-β | Teriflunomide 7 mg + IFN-β | Teriflunomide 14 mg + IFN-β | Placebo + GA | Teriflunomide 7 mg + GA | Teriflunomide 14 mg + GA
Number analyzed (Participants) | 41 | 37 | 38 | 41 | 42 | 40
percent probability
  Probability of disability progression at 24 weeks | 0.0 [0.0 to 0.0] | 3.0 [0.0 to 8.9] | 2.7 [0.0 to 7.9] | 2.5 [0.0 to 7.3] | 0.0 [0.0 to 0.0] | 5.6 [0.0 to 13.2]
  Probability of disability progression at 48 weeks | 0.0 [0.0 to 0.0] | 11.1 [0.0 to 23.1] | 6.4 [0.0 to 15.2] | 10.6 [0.7 to 20.4] | 3.3 [0.0 to 9.8] | 12.8 [1.0 to 24.6]

6. Secondary Outcome: Cerebral Magnetic Resonance Imaging [MRI] Assessment: Change From Baseline in Total Lesion Volume (Burden of Disease)
Description: Total lesion volume is the sum of the total volume of all T2-lesions and the total volume all T1-hypointense post-gadolinium lesions measured through T2/proton density scan analysis and gadolinium-enhanced T1 scan analysis.
  Least-square means were estimated using two Mixed-effect models with repeated measures [MMRM] on cubic root transformed volume data:
  * Model 1 (IFN-β groups): treatment group, region of enrollment, IFN-β dose level, visit, treatment-by-visit interaction, baseline value (cubic root transformed), and baseline-by-visit interaction as factors;
  * Model 2 (GA groups): treatment group, region of enrollment, visit, treatment-by-visit interaction, baseline value (cubic root transformed), and baseline-by-visit interaction as factors.
Time Frame: baseline (before randomization in PDY6045 or PDY6046) and 48 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mililiters (mL)
Arm/Group | Placebo + IFN-β | Teriflunomide 7 mg + IFN-β | Teriflunomide 14 mg + IFN-β | Placebo + GA | Teriflunomide 7 mg + GA | Teriflunomide 14 mg + GA
Number analyzed (Participants) | 41 | 37 | 38 | 41 | 42 | 40
mililiters (mL) | -0.017 (0.028) [-11.29 to 7.26] | -0.011 (0.030) [-9.63 to 3.35] | -0.012 (0.029) [-8.97 to 7.29] | 0.016 (0.036) [-15.62 to 19.44] | -0.010 (0.037) [-15.91 to 7.04] | -0.063 (0.039) [-10.69 to 7.02]

7. Secondary Outcome: Cerebral MRI Assessment: Number of Gd-enhancing T1-lesions Per Scan (Poisson Regression Estimates)
Description: Number of Gd-enhancing T1-lesions per scan is obtained from the total number of Gd-enhancing T1-lesions observed during the study divided by the total number of scans performed during the study.
  To account for the different number of scans among participants, two Poisson regression models with robust error variance were used (total number of Gd-enhancing T1-lesions as response variable, log-transformed number of scans as "offset" variable and:
  * Model 1 (IFN-β groups): Treatment group, region of enrollment, IFN-β dose level and baseline number of Gd-enhancing T1-lesions as covariates
  * Model 2 (GA groups): Treatment group, region of enrollment and baseline number of Gd-enhancing T1-lesions as covariates)
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: lesions per scan
Arm/Group | Placebo + IFN-β | Teriflunomide 7 mg + IFN-β | Teriflunomide 14 mg + IFN-β | Placebo + GA | Teriflunomide 7 mg + GA | Teriflunomide 14 mg + GA
Number analyzed (Participants) | 41 | 37 | 38 | 41 | 42 | 40
lesions per scan | 0.521 [0.318 to 0.854] | 0.080 [0.032 to 0.204] | 0.090 [0.052 to 0.154] | 0.333 [0.171 to 0.649] | 0.120 [0.059 to 0.243] | 0.178 [0.098 to 0.324]

8. Primary Outcome: Liver Function: Number of Participants With Potentially Clinically Significant Abnormalities [PCSA]
Description: PCSA values are abnormal values considered medically important by the Sponsor according to predefined criteria based on literature review.
  Hepatic parameters thresholds were defined as follows:
  * Alanine Aminotransferase [ALT] >3, 5, 10 or 20 Upper Normal Limit [ULN];
  * Aspartate aminotransferase [AST] >3, 5, 10 or 20 ULN;
  * Alkaline Phosphatase >1.5 ULN;
  * Total Bilirubin [TB] >1.5 or 2 ULN;
  * ALT >3 ULN and TB >2 ULN;
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo + IFN-β | Teriflunomide 7 mg + IFN-β | Teriflunomide 14 mg + IFN-β | Placebo + GA | Teriflunomide 7 mg + GA | Teriflunomide 14 mg + GA
Number analyzed (Participants) | 41 | 37 | 38 | 40 | 42 | 41
participants
  ALT >3 ULN | 2 | 1 | 3 | 1 | 0 | 1
  - ALT >5 ULN | 1 | 0 | 1 | 1 | 0 | 1
  - ALT >10 ULN | 0 | 0 | 0 | 1 | 0 | 0
  AST >3 ULN | 1 | 0 | 1 | 1 | 0 | 0
  - AST >5 ULN | 1 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase >1.5 ULN | 1 | 0 | 0 | 0 | 0 | 0
  TB >1.5 ULN | 0 | 0 | 0 | 0 | 0 | 0
  ALT >3 ULN and TB >2 ULN | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Cerebral MRI Assessment: Total Volume of Gd-enhancing T1-lesions Per Scan
Description: Total volume of Gd-enhancing T1-lesions per scan is obtained from the sum of the volumes of Gd-enhancing T1-lesions observed during the study divided by the total number of scans performed during the study.
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Number; unit: mililiters per scan
Arm/Group | Placebo + IFN-β | Teriflunomide 7 mg + IFN-β | Teriflunomide 14 mg + IFN-β | Placebo + GA | Teriflunomide 7 mg + GA | Teriflunomide 14 mg + GA
Number analyzed (Participants) | 41 | 37 | 38 | 41 | 42 | 40
mililiters per scan | 0.068 | 0.019 | 0.020 | 0.052 | 0.031 | 0.014

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected regardless of seriousness or relationship to the drug, spanning from signature of the Informed Consent up to the last visit.
Description: The analysis was performed on the exposed population and included all AE that developed or worsened from first study drug intake in PDY6045/PDY6046 study up to 112 days after last intake in initial study or in the extension study, whichever occured first (64 weeks max).
Arm/Group | Placebo + IFN-β | Teriflunomide 7 mg + IFN-β | Teriflunomide 14 mg + IFN-β | Placebo + GA | Teriflunomide 7 mg + GA | Teriflunomide 14 mg + GA
Serious Adverse Events (participants affected / at risk) | 2/41 | 4/37 | 1/38 | 6/40 | 5/42 | 2/41
Other Adverse Events (participants affected / at risk) | 28/41 | 33/37 | 32/38 | 34/40 | 30/42 | 34/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + IFN-β (N=41) | Teriflunomide 7 mg + IFN-β (N=37) | Teriflunomide 14 mg + IFN-β (N=38) | Placebo + GA (N=40) | Teriflunomide 7 mg + GA (N=42) | Teriflunomide 14 mg + GA (N=41)
Abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Mastoiditis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasticity (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 0 | 2 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + IFN-β (N=41) | Teriflunomide 7 mg + IFN-β (N=37) | Teriflunomide 14 mg + IFN-β (N=38) | Placebo + GA (N=40) | Teriflunomide 7 mg + GA (N=42) | Teriflunomide 14 mg + GA (N=41)
Bronchitis (Infections and infestations) | 0 | 1 | 2 | 1 | 3 | 2
Ear infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 3 | 0 | 0
Influenza (Infections and infestations) | 3 | 1 | 0 | 1 | 1 | 2
Nasopharyngitis (Infections and infestations) | 3 | 3 | 5 | 6 | 7 | 4
Respiratory tract infection (Infections and infestations) | 2 | 2 | 0 | 0 | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 5 | 2 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 2 | 0 | 1 | 4
Upper respiratory tract infection (Infections and infestations) | 4 | 2 | 2 | 6 | 2 | 4
Urinary tract infection (Infections and infestations) | 7 | 4 | 1 | 6 | 5 | 4
Anxiety (Psychiatric disorders) | 1 | 2 | 1 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 1 | 2 | 5 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 3 | 1 | 1 | 3
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 3
Dizziness (Nervous system disorders) | 2 | 0 | 1 | 3 | 1 | 1
Headache (Nervous system disorders) | 2 | 2 | 6 | 7 | 6 | 7
Hypoaesthesia (Nervous system disorders) | 2 | 0 | 2 | 2 | 2 | 2
Muscle spasticity (Nervous system disorders) | 0 | 0 | 0 | 0 | 4 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 3
Sciatica (Nervous system disorders) | 0 | 2 | 1 | 2 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 0 | 3 | 1 | 0
Hypertension (Vascular disorders) | 1 | 3 | 4 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2 | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1 | 3 | 2 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 4
Diarrhoea (Gastrointestinal disorders) | 6 | 4 | 4 | 2 | 3 | 8
Nausea (Gastrointestinal disorders) | 3 | 0 | 5 | 3 | 5 | 5
Vomiting (Gastrointestinal disorders) | 2 | 1 | 4 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 3 | 3 | 1 | 5 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 3 | 6
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 2 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 4 | 2 | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 4 | 3 | 2
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 3 | 3
Asthenia (General disorders) | 1 | 1 | 3 | 0 | 0 | 1
Fatigue (General disorders) | 4 | 2 | 5 | 7 | 4 | 7
Oedema peripheral (General disorders) | 1 | 0 | 0 | 3 | 2 | 2
Alanine aminotransferase increased (Investigations) | 6 | 7 | 12 | 2 | 3 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 7 | 4 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 3 | 1 | 1 | 1 | 0
Blood pressure increased (Investigations) | 0 | 1 | 3 | 0 | 0 | 1
Blood triglycerides increased (Investigations) | 1 | 1 | 2 | 1 | 1 | 0
Lipase increased (Investigations) | 0 | 0 | 2 | 1 | 0 | 3
Lymphocyte count decreased (Investigations) | 1 | 4 | 5 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 1 | 4 | 0 | 1 | 1
Protein urine present (Investigations) | 3 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 3 | 3 | 4 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 1 | 1 | 2
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months after trial completion, the Investigator can publish the results. Prior to publication, the sponsor shall review the manuscript and can request changes, provided they do not jeopardize the accuracy and/or the scientific value of the publication. The approval is given in writing by the sponsor, not exceeding 90 days.

To protect by property right the sponsor can postpone the publication of any information, for a period not exceeding 18 months.